CLINICAL TRIAL: NCT01189851
Title: Intraoperative Radiotherapy (IORT) for the Management of Carcinoma of the Breast: Use of Mammography, Ultrasonography,and Contrast-Enhanced Magnetic Resonance Imaging (CE-MRI) to Identify Candidates for IORT
Brief Title: Intraoperative Radiotherapy for Early Stage Breast Cancer
Acronym: IORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IORT
Record Dates: First submitted 2010-06-21; First posted 2010-08-27 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: breast; IORT; electronic brachytherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IORT (Other): Treated with Intraoperative Radiation Therapy
  Interventions: Device: Intraoperative Radiotherapy

INTERVENTIONS:
Device: Intraoperative Radiotherapy — The Axxent eBx™ System utilizes a miniaturized high dose rate (HDR) X-ray source to apply radiation directly to the cancerous tumor bed and provides brachytherapy when the physician chooses to deliver intracavitary or interstitial radiation to the surgical margins following lumpectomy for breast cancer.
  Other Names: 510(k) Number K050843; Axxent™ Electronic Brachytherapy System

SUMMARY:
Up to 200 patients with biopsy proven early stage breast cancer selecting Wide Local Excision (WLE) will undergo mammography, ultrasound (of affected breast and ipsilateral axilla) and contrast enhanced-magnetic resonance imaging (CE-MRI) of the affected breast to evaluate the extent of disease.

DETAILED DESCRIPTION:
Patients will be deemed eligible for immediate IORT if the invasive cancer lesion is estimated to measure ≤ 3.0 centimeters maximum dimension by mammogram, ultrasound, and CE-MRI and is thought to be resectable with WLE and clear surgical margins, with clinically staged N0M0 disease, minimum age of 48, and histology of invasive ductal or lobular carcinoma of the breast. The lesion size determined by imaging will be compared with lesion size and surgical margin status obtained from the surgical pathology specimen to evaluate the ability of mammography combined with ultrasound and CE-MRI to identify suitable candidates for immediate IORT.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent. Each eligible patient must willingly give written consent after being informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts.
2. Histology. Patients must have biopsy-proven invasive ductal or lobular carcinoma of the breast.
3. Female, age ≥ 48 years.
4. Clinically and/or histologically negative axillary lymph nodes.
5. No imaging or clinical findings that indicate metastatic disease.
6. Procedure deemed appropriate based upon factors such as breast size by the treating surgeon and radiation oncologist.

Exclusion Criteria:

1. Male sex
2. Age < 48
3. Non-epithelial breast malignancies such as sarcoma, lymphoma, or metastatic breast cancer
4. Pregnancy or lactation
5. Serious psychiatric or addictive disorders
6. More than one obvious cancer in the same breast as diagnosed by clinical examination, mammography, ultrasonography, and/or CE-MRI.
7. Bilateral breast cancer at the time of diagnosis, unless agreed upon by the surgeon and radiation oncologist.
8. Ipsilateral breast with a previous cancer and/or irradiation.
9. Extensive Intraductal Component (DCIS ≥ 25% of the tumor).
10. Patients presenting with gross nodal disease considered to be clinically malignant by scanning or proven cytologically or by sentinel node biopsy will be cancelled.
11. Previous history of malignant disease does not preclude entry if the expectation of relapse-free survival at 10 years is 90% or greater.
12. Lymphovascular invasion on needle biopsy.
13. Patients undergoing primary medical treatment (hormones or chemotherapy) as initial treatment with intent to reduce tumor size.

Min Age: 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-06 (Actual); Primary Completion 2023-09 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants Receiving Additional Surgery Because of Positive or Close Margins as a Measure of the Accuracy of Pre-Operative Assessment | 10 years
  Invasive cancer margins <1 mm and/or non-invasive cancer margins < 2 mm are considered close or positive. Approximately 15% of patients treated with IORT have close or positive margins on pathologic assessment following IORT therapy and are recommended for additional therapy including re-excision, whole breast radiation or both.

SECONDARY OUTCOMES:
Proportion of Participants Recommended to Have Additional Whole Breast Radiation Therapy (WBRT) Because of High Risk Features Found on Final Pathology as a Measure of the Accuracy of Pre-Operative Assessment | 5 years
  Patients treated with IORT that have high risk features on final pathologic exam, including close/positive margins, tumor size >30 mm, positive lymph nodes and lympho-vascular invasion (LVI) are recommended for additional therapy including re-excision, whole breast radiation or both.
Proportion of Participants with Tumor Size Larger than the Entry Criteria Size and/or Positive Lymph Nodes as a Measure of the Accuracy of Pre-Operative Assessment | 5 years
  Both tumor size and lymph node status are estimated prior to surgery using mammography, ultrasound and MRI (unless excluded for medical reasons). Patients with estimated tumor spans > 30 mm or positive lymph nodes are excluded from IORT.
Proportion of Participants with Serious Adverse Events and/or Complications as a Measure of the Safety of the Treatment Algorithm | 5 years
  We will be monitoring acute side effects attributed directly to IORT. These includ erythemia, hyperpigmentation, fibrosis, seromas, infection and wound breakdown.
Cosmesis Scores by Physician and Self-Assessment | 5 years
  The first 213 IORT patients treated will be asked to fill out a yearly cosmesis assessment. Patients filled out these assessments for an average of 2-3 years.
Progression Free Survival in the First Five Years | 5 years
  We will follow progression free survival for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter V Chen, MD, Principal Investigator — Hoag Memorial Hospital Presbyterian
Locations (1):
- Hoag Memorial Hospital Presbyterian - Cancer Center, Newport Beach, California, United States